CLINICAL TRIAL: NCT00459238
Title: A Telephone-Based Education and Prevention Intervention for Teens and Young Adults
Brief Title: Telephone-Based Cancer Education With or Without Telephone-Based Counseling in Young Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDR0000538178; R03CA119686 (NIH); P30CA051008 (NIH); GUMC-2006-243
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-02

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Counseling; Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: counseling intervention — subjects will receive telephone based counseling
Other: educational intervention — subjects will received telephone based education

SUMMARY:
RATIONALE: Telephone-based cancer education and counseling may help participants learn about ways of preventing cancer and choose a lifestyle that will help them stay healthy as they grow older.

PURPOSE: This randomized clinical trial is studying telephone-based cancer education and telephone-based counseling to see how well they work compared with telephone-based cancer education alone in young participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of telephone-based cancer education with vs without counseling in younger participants.

Secondary

* Determine the mechanisms by which education with counseling may impact cancer-relevant cognitive and behavioral outcomes.
* Identify teens who may be most and least likely to benefit from education with counseling.

OUTLINE: This is a pilot, controlled, randomized study. Participants are stratified according to age (13-14 years vs 15 years vs 16 years vs 17 years vs 18-21 years), gender, race (white vs black vs other), and health status (chronic disease vs no chronic disease). Participants are randomized to 1 of 2 education arms.

* Arm I: Participants undergo cancer education sessions via telephone over 45 minutes once a week for 8 weeks.
* Arm II: Participants under cancer education sessions as in arm I and counseling techniques during the same telephone sessions.

In both arms, participants receive an intervention kit by mail before the first telephone call. The intervention kit includes age-appropriate self-help materials.

PROJECTED ACCRUAL: A total of 300 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* No life-threatening illness (e.g., cancer)

  * Chronic illnesses (e.g., asthma, diabetes) allowed with permission by physician

PATIENT CHARACTERISTICS:

* No serious restrictions on physical activity, diet, or nutrition, including any of the following:

  * Untreated exercise-induced asthma
  * Orthopedic or neurological problems
  * Medical conditions affecting nutritional status, intestinal absorption, or response to nutritional intervention (e.g., inflammatory bowel disease)
* No serious mental illness or developmental disability that would preclude study compliance, including eating disorders
* Must adequately understand, speak, and read English

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Multiple risk factor index | 6 months
Knowledge | 6 months
Health history taking | 3 months
Nutrition | 6 months
Physical activity | 6 months
Tobacco use intentions and behavior | 6 months
Alcohol use intentions and behavior | 6 months
Screening intentions | 6 months
Self-efficacy | 6 months
Perceived benefits | 6 months
Perceived barriers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Tercyak, PhD, Study Chair — Lombardi Comprehensive Cancer Center
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia, United States